CLINICAL TRIAL: NCT03415256
Title: The Effects of Passive Vibration in Patients With Diabetic Peripheral Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of time currently.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Everett Lohman, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5170453
Record Dates: First submitted 2017-12-12; First posted 2018-01-30 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: * After completing the tests, you will be randomly assigned by the computer to either the treatment group or control group.
  * The treatment group will receive a passive vibration treatment for 15 minutes twice a week for 4 weeks.
  * The control group will not receive any treatment and they will continue their usual lifestyle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- passive vibration group (Experimental): The passive vibration group patients will receive passive vibration (50 Hz, one cycle= 60 seconds working time with 2 seconds rest time) on their calf in supine position for ten minutes. The total number of sessions will be nine. Passive vibration will be given to the treatment group twice a week for four weeks (eight sessions) and the ninth session will be the follow up. At every session, the skin blood flow will be measured before, immediately, and 15 minutes after passive vibration.
  Interventions: Other: passive vibration
- no passive vibration group (Active Comparator): The control group will not receive any treatment and continue their usual lifestyle. Balance, sensory measurement and skin blood flow will be taken at the beginning of the study, prior to the 5th treatment, and 1 week after the last intervention .
  Interventions: Other: no passive vibration

INTERVENTIONS:
Other: passive vibration — The passive vibration is delivered using a Physio Plate (Domino S.R.L, San Vendemiano, Italy). The frequency delivered is 50 Hz for a total number of ten cycles for a period of ten minutes approximately (one cycle= 60seconds working time with 2 seconds rest time).
  Arms: passive vibration group
Other: no passive vibration — The control group will not receive any treatment and continue their usual lifestyle.
  Arms: no passive vibration group

SUMMARY:
The purpose of this study is to examine the effects of passive vibration (PV) in improving balance and sensation in patients with diabetic peripheral neuropathy (DPN).

DETAILED DESCRIPTION:
The study involves the following:

* Visit 1:
* Particpant's age, height, gender, and weight will be collected.
* Participant will fill out a questionnaire to assess participant's nerve function. This process will take approximately 2.5 minutes.
* Investigator will measure participant's balance, sensation, and skin blood flow (SBF).
* After completing the tests, participant will be randomly assigned by the computer to either the treatment group or control group.
* The treatment group will receive a passive vibration treatment for 15 minutes twice a week for 4 weeks.
* The control group will not receive any treatment and they will continue their usual lifestyle.
* Visit 2 through 8:
* The treatment group will receive a passive vibration for 15 minutes followed by SBF measurement.
* The control group will continue their usual lifestyle.
* In the fifth session, the treatment and control groups will come back for tests.
* Visit 9 (follow-up):

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Diabetic Peripheral Neuropathy
* Minimum age 40 years
* Maximum Age 75 years
* Ability to stand for a minimum of five minutes

Exclusion Criteria:

* Neurological Disorders
* Bleeding Disorders
* Leg Ulcers
* Cardiovascular Diseases
* Complete absence of sensation in lower extremities (i.e. 6.65 in monofilament test)
* Self-reported pregnancy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Skin blood flow | Change between Baseline and Week Nine Visit
  Patient will be positioned in prone on a plinth as their skin is marked for blood flow assessment. A 3 cm x 3 cm square shape will be marked on the posterior aspect of the calf (muscle belly) and on the plantar aspect of the first three metatarsal heads. MOOR Full-field Laser Perfusion Image(FLPI) (MOOR FLPI V 2.1, Oxford, England) will be used for measurement of skin blood flow in a patient with DPN, which will be pre-warmed for about 30 minutes. The perpendicular red light laser beam will be used to capture SBF and blood flow is measured in '"Flux" unit.

SECONDARY OUTCOMES:
balance | at each of the nine visits( 90 minutes each visit: twice per week)
  The NeuroCom Smart Balance Master System Computerized dynamic posturography (CDP) will be used in this research to measure balance. The platform consists of two force plates that can be modulated in the up-down and anterior-posterior direction. The sensory organization test (SOT) will be used to measure balance. The result of CDP determines any anomalies in visual, somatosensory and vestibular systems that control posture.

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, DSc, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No